CLINICAL TRIAL: NCT01331902
Title: Comparison of Hyperemic Efficacy Between Nicorandil and Adenosine for Fractional Flow Reserve (FFR) Measurement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Boramae Hospital (Other); Inje University Ilsan Paik Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Bon- Kwon Koo / prof, Cardiovascular Center, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1101-069-348
Record Dates: First submitted 2011-04-01; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Adenosine; Nicorandil; Fractional Flow Reserve; Maximal Hyperemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adenosine Followed by Nicorandil (Experimental)
  Interventions: Other: Maximal Hyperemia with Adenosine Followed by Nicorandil
- Nicorandil Followed by Adenosine (Experimental)
  Interventions: Other: Maximal Hyperemia with Nicorandil Followed by Adenosine

INTERVENTIONS:
Other: Maximal Hyperemia with Adenosine Followed by Nicorandil — Firstly FFR was measured with intravenous adenosine infusion (140 μg•min-1•kg-1) via femoral vein or antecubital vein. Secondly with intracoronary adenosine bolus injection (80μg, 40μg to LCA and RCA, respectively). Lastly with intracoronary nicorandil bolus injection (1mg followed by 2mg).
  Arms: Adenosine Followed by Nicorandil
Other: Maximal Hyperemia with Nicorandil Followed by Adenosine — Firstly FFR was measured with intracoronary nicorandil bolus injection (1mg followed by 2mg). Secondly with intravenous adenosine infusion (140 μg•min-1•kg-1) via femoral vein or antecubital vein. Lastly with intracoronary adenosine bolus injection (80μg, 40μg to LCA and RCA, respectively).
  Arms: Nicorandil Followed by Adenosine

SUMMARY:
The purpose of this study is to evaluate the efficacy of nicorandil in the achievement of maximal coronary hyperemia compared with adenosine.

ELIGIBILITY:
Inclusion Criteria:

* non -infarct related, patients with moderate coronary artery stenosis
* normal left ventricular ejection fraction on echocardiogram

Exclusion Criteria:

* infarct-related arteries or clinically unstable state
* collateral blood flow to the target vessel is shown
* atrioventricular block on electrocardiogram
* reduced left ventricular ejection fraction (<50%) or left ventricular hypertrophy on echocardiogram
* contraindication of adenosine
* bronchial asthma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Fractional Flow Reserve at Maximal Hyperemia | 1 day

SECONDARY OUTCOMES:
Time to Maximal Hyperemia | 1 day
Changes in Heart Rate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD. PhD, Study Chair — Department of Internal Medicine, Cardiovascular Center, Seoul National University Hospital
Locations (1):
- Cardiovascular Center, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jang HJ, Koo BK, Lee HS, Park JB, Kim JH, Seo MK, Yang HM, Park KW, Nam CW, Doh JH, Kim HS. Safety and efficacy of a novel hyperaemic agent, intracoronary nicorandil, for invasive physiological assessments in the cardiac catheterization laboratory. Eur Heart J. 2013 Jul;34(27):2055-62. doi: 10.1093/eurheartj/eht040. Epub 2013 Feb 8. PMID 23396491